CLINICAL TRIAL: NCT03240484
Title: Examining Effects of Spinal Arthrodesis on Outcomes Following Total Hip Arthroplasty
Brief Title: Examining Effects of Spinal Fusion on Outcomes Following Total Hip Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Wade Gofton, Orthopaedic Surgeon, Ottawa Hospital Research Institute
Other Study IDs: 20170312
Record Dates: First submitted 2017-07-21; First posted 2017-08-07 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Spinal Fusion; Total Hip Replacement
MeSH Terms: interventions — Diagnostic Imaging; Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Spine Fusion and Total Hip Replacement: Any patient who has undergone spine fusion (SF) and total hip arthroplasty (THA). Patients will undergo x-ray imaging and complete functional assessment questionnaires. Patients may additionally be asked to participate in a gait analysis in a Human Movement Laboratory.
  Interventions: Diagnostic Test: X-Ray Imaging; Other: Gait Analysis
- Total Hip Replacement Group: Any patient who has had THA only (no spine fusion surgery). Patients will undergo x-ray imaging and complete functional assessment questionnaires. Patients may additionally be asked to participate in a gait analysis in a Human Movement Laboratory.
  Interventions: Diagnostic Test: X-Ray Imaging; Other: Gait Analysis
- Spine Fusion Only Group: Any patient who has had spine fusion only (no hip replacement surgery). Patients will undergo x-ray imaging and complete functional assessment questionnaires.
  Interventions: Diagnostic Test: X-Ray Imaging

INTERVENTIONS:
Diagnostic Test: X-Ray Imaging — X-Ray imaging in the following positions: Lateral standing, lateral seated, standard standing AP pelvis and AP pelvis lying down.
Other: Gait Analysis — Certain patients may be asked to participate in a motion analysis procedure at the Human Movement Laboratory at the University of Ottawa. This procedure takes approximately 1.5 hours and you will only be asked to participate in the motion analysis procedure once. Participants will change into a custom-designed tight body suit, which has reflective markers on its surface for infrared video capture. Participants will then have pairs of surface electromyography (EMG) electrodes placed on certain areas of the skin on the legs and on the back. Wearing the EMG electrodes and marker suit, participants will perform 5 trials of walking on a level walkway, walking up and down a 3-step staircase, sitting from a standing position, and standing from a seated position.
  Groups: Spine Fusion and Total Hip Replacement; Total Hip Replacement Group

SUMMARY:
The purpose of the study is to explore the long term functional status of people who have had both a spinal fusion procedure and a total hip replacement.

DETAILED DESCRIPTION:
The purpose of the study is to explore the long term functional status of people who have had both a spinal fusion procedure and a total hip replacement. Studies have found that those who have received spinal fusion may have worse outcomes following a total hip replacement than those who have not received a spinal fusion. The information obtained from this study will allow surgeons and researchers to better understand why some who've had a spine fusion have more complications post total hip replacement compared to those who did not have spinal fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* Willing to come to the Civic Campus for a surgical follow-up visit
* Speaks English and/or French
* Group 1 patients must have had a spine fusion (SF) and total hip arthroplasty (THA)
* Group 2 patients must have had a total hip replacement (THA) and no history of spine fusion (SF)
* Group 3 patients must have had a spine fusion (SF) and no history of total hip arthroplasty (THA)

Exclusion Criteria:

* Patient does not meet all 'inclusion' criteria
* Patient is unable to answer questionnaires
* Unable to get x-rays for other medical reasons
* Severe dementia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 70 patients who underwent total hip arthroplasty (THA) and spine fusion (SF) surgery will be called by the surgeon or research team and asked if they wish to participate in the study. A second group of approximately 45 patients who have only had a THA (and no SF) will serve as a comparison group. A third group of approximately 45 patients who have only had an SF surgery (and no THA) will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Implant positioning | 6months or greater post-operative
  Radiographic assessment (x-ray cup orientation measurements)

SECONDARY OUTCOMES:
Hip dysfunction and osteoarthritis outcome score (HOOS) | 6months or greater post-operative
  Disease-specific quality of life measure
Oxford Hip Score | 6months or greater post-operative
  Disease-specific quality of life measure
SF-12 Questionnaire | 6months or greater post-operative
  Patient-reported overall quality of life measure
Oswestry low back disability questionnaire | 6months or greater post-operative
  Assessment of low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Wade Gofton, MD, FRCSC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No